CLINICAL TRIAL: NCT00154115
Title: Efficacy of Levosimendan in Cardiac Failure After Heart Valve Surgery
Brief Title: Levosimendan in High Risk Heart Valve Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Pasi Lahtinen, MD, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KUH5070178; 106/2004
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Heart Failure
Keywords: heart failure; levosimendan; cardiac surgery
MeSH Terms: conditions — Heart Failure | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Levosimendan
  Interventions: Drug: levosimendan
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: levosimendan — Intravenous infusion, blus 24 mcg/kg in 30-minutes followed by 0.2 mcg/kg/min up to 24 hours
  Arms: 1
Drug: placebo — Placebo
  Arms: 2

SUMMARY:
Prospective, randomized, double blind study investigating the efficacy of levosimendan in heart failure after cardiac surgery.

Study hypothesis: Levosimendan diminishes the need for adrenergic inotropic drugs and morbidity and may improve survival after heart valve surgery.

DETAILED DESCRIPTION:
200 patients are prospectively randomized in a double blind study investigating the efficacy of levosimendan in heart failure after cardiac surgery. Levosimendan/placebo is administered as 24 hour continuous infusion beginning after anesthesia induction. Primary endpoint being adrenergic inotrope need after cardiopulmonary bypass and secondary endpoints hospital and 6-month mortality and major organ failure.

ELIGIBILITY:
Inclusion Criteria:

Eligible for cardiac valve or combined CABG and cardiac valve surgery:

* Clinical signs of cardiac insufficiency

Exclusion Criteria:

* Endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Heart failure necessitating inotropic drug administering after heart valve surgery | Postoperative hospital period

SECONDARY OUTCOMES:
Hospital morbidity and mortality | Postoperative hospital period
Postoperative mortality at six months | Six months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Pasi K Lahtinen, MD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland